CLINICAL TRIAL: NCT03705273
Title: Comparison of Dexamethasone Oral Preparations to Assess Palatability and Adverse Effects in Children With Asthma and Croup
Brief Title: Comparison of Dexamethasone Oral Preparations to Assess Taste and Acceptance in Children With Asthma and Croup
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Dr. Arnold assisted in designing and initiating study for a pharmacology PhD candidate. The candidate left the institution and study enrollment was terminated.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Donald H Arnold, Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181682
Record Dates: First submitted 2018-10-09; First posted 2018-10-15 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Asthma; Croup
MeSH Terms: conditions — Asthma; Croup | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone IV for PO (Experimental): Dexamethasone IV for PO solution mixed with sugar syrup to be given orally
  Interventions: Drug: Dexamethasone IV for PO
- Dexamethasone crushed tablets (Active Comparator): Dexamethasone tablet crushed and placed in apple sauce or pudding to be given orally
  Interventions: Drug: Dexamethasone crushed tablets

INTERVENTIONS:
Drug: Dexamethasone IV for PO — Common pediatric emergency department practice
  Other Names: Dexamethasone injection
  Arms: Dexamethasone IV for PO
Drug: Dexamethasone crushed tablets — Alternative route of administration for patients unable to swallow tablet whole
  Other Names: Dexamethasone oral tablet
  Arms: Dexamethasone crushed tablets

SUMMARY:
Study of the palatability and acceptability of dexamethasone oral tablets crushed and placed in apple sauce or pudding in comparison with the IV solution mixed with sugar syrup and given orally. It is hypothesized that dexamethasone tablets crushed and administered in apple sauce or pudding will be more palatable and acceptable for pediatric patients receiving dexamethasone for an acute asthma exacerbation or croup.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute asthma exacerbation or croup (laryngotracheitis) in the Vanderbilt Children's Hospital Emergency Department
* Age 1 to 7 years
* Dexamethasone treatment indicated
* No other acute or chronic process accounting for signs and symptoms (e.g., foreign body aspiration, pneumonia, cystic fibrosis)
* Have not received systemic corticosteroid for current episode prior to enrollment

Exclusion Criteria:

* Allergy to dexamethasone or apple sauce and pudding
* Unable to take medication orally

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Arnold, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goettel AM, Hanson HR, Overfield J, Thornton C, Arnold DH. Tastes great, less filling! Randomized trial comparing perceived palatability of dexamethasone preparations in children. Ann Allergy Asthma Immunol. 2023 Jan;130(1):114-115. doi: 10.1016/j.anai.2022.09.016. No abstract available. PMID 36596609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty participants were enrolled and randomized, of which 20 were randomized to receive dexamethasone tablets.
Groups:
- Dexamethasone Tablets: Dexamethasone tablets crushed and administered in apple sauce or pudding at a dose of 0.6 mg/kg
- Dexamethasone-IV Solution-in-syrup: Dexamethasone-IV solution-in-syrup at a dose of 0.6 mg/kg
Period: Overall Study
Arm/Group | Dexamethasone Tablets | Dexamethasone-IV Solution-in-syrup
Started | 20 (Planned enrollment of 110 participants in the arm was not achieved due to lack of study personnel.) | 20 (Planned enrollment of 110 participants in the arm was not achieved due to lack of study personnel.)
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexamethasone Crushed Tablets: Dexamethasone tablet crushed and placed in apple sauce or pudding to be given orally or dexamethasone IV solution in cherry syrup
- Total: Total of all reporting groups
Arm/Group | Dexamethasone IV for PO | Dexamethasone Crushed Tablets | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.75 (1.88) | 2.70 (1.92) | 2.75 (1.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 13 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Diagnosis asthma [Count of Participants; unit: Participants] | 15 | 16 | 31
Diagnosis croup [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nausea
Description: Presence of nausea after medication administration (yes/no) measured by participant self-report
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Groups:
- Dexamethasone Tablets: Dexamethasone tablets crushed and mixed in apple sauce
- Dexamethasone IV for PO: Dexamethasone IV solution mixed with cherry syrup
Arm/Group | Dexamethasone Tablets | Dexamethasone IV for PO
Number analyzed (Participants) | 20 | 20
Participants | 3 | 0

2. Secondary Outcome: Number of Participants Requiring Second Dose of Dexamethasone
Description: Reason for patient needing a second dose of dexamethasone; such as spit dose up or vomiting dose
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Tablets | Dexamethasone IV for PO
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Time of randomization up to one hour after last dose of treatment
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Dexamethasone IV for PO | Dexamethasone Crushed Tablets
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03705273/Prot_SAP_000.pdf